CLINICAL TRIAL: NCT03073876
Title: Detecting an Early Response to Donepezil With Measures of Visual Attention
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Collaborators: Queens College, The City University of New York (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Other
Other Study IDs: WUH 05030
Record Dates: First submitted 2017-02-15; First posted 2017-03-08 (Actual); Results first posted 2019-11-05 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-01

CONDITIONS: Alzheimer Disease
Keywords: Alzheimer Disease; Attention; Donepezil hydrochloride
MeSH Terms: conditions — Alzheimer Disease | interventions — Donepezil

STUDY DESIGN:
Intervention Model Description: Double Blind Placebo Control
Who Masked: Participant, Care Provider, Investigator
Masking Description: Study drug was prepared by research pharmacist who was the only person privy to group assignment. Drug and Placebo pills looked identical.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Drug (Experimental): Participants in the Drug group received oral 5mg of Donepezil Hydrochloride daily for 6 months. The Drug group was assessed at baseline, after approximately 6 weeks and after 6 months of treatment. The baseline to 6 weeks phase was part of the double-blind, placebo controlled portion of the trial.
  Interventions: Drug: Donepezil Hydrochloride
- Placebo (Placebo Comparator): Participants in the placebo group first received oral administration of a placebo pill for approximately 6 weeks. After that initial interval, the study was unblinded and participants in the placebo group then received 5mg of donepezil hydrochloride treatment for 6 months.
  The Placebo group was evaluated at baseline, after 6 weeks of placebo, after 6 weeks of donepezil hydrochloride drug treatment, and 6 months of donepezil hydrochloride treatment.
  Interventions: Drug: Donepezil Hydrochloride; Drug: Placebo

INTERVENTIONS:
Drug: Donepezil Hydrochloride — 5mg of Donepezil Hydrochloride by mouth
  Other Names: Aricept
Drug: Placebo — prepared placebo looking exactly the same as drug. Participants took placebo by mouth for approximately 6 weeks, and after unblinding, they took donepezil hydrochloride for 6 months.
  Other Names: Placebo pill
  Arms: Placebo

SUMMARY:
Acetylcholinesterase inhibitors (AChE-I) comprise a class of drugs used to treat Alzheimer's disease (AD), but controversy about their usefulness remains. Modest response rates of treated versus placebo groups, small effect sizes with respect to efficacy, drug costs, and clinical relevance of the effects are problematic. Standard efficacy measures of efficacy are not sufficiently sensitive, and trying to assess cognitive change after 4-6 months of therapy confounds the drug effect and the natural progression of the disease.

Surprisingly, attention has never been included in the assessment of AChE-I drugs. The rationale for using attentional measures are that (1) Attentional deficits are recognized as a critical cognitive change in the earliest phases of AD; (2) Attentional function is directly mediated by the cholinergic system, and responds rapidly to cholinergic augmentation, particularly on tasks that tax available attentional capacity are dose dependent; and (3) Acetylcholine is depleted in AD. However, the link between attention and cholinergic depletion in AD has not been fully explored, especially with regard to response to cholinergic treatment.

The study tests if attentional performance can be a more sensitive marker of response. In a longitudinal study we measure attentional, as well as cognitive and behavioral performance in de novo AD patients undergoing donepezil treatment. The investigators develop visual attentional measures and contrast them to global and domain-specific cognitive scores on three occasions (T1) baseline pre-treatment, (T2) after approximately 6 weeks, and (T3) after 6 months treatment. The T1-to-T2 arm is a double-blind placebo control period, after which members of the placebo group start open-label treatment. The assessment at 6 months allows us to determine whether the changes seen earlier at T2 can predict patients who respond, or determine which measures best predict response.

We hypothesize that attention measures are more sensitive than standard global measures or other cognitive domains and that the change of attentional function can be detected after only after approximately 6 weeks treatment.

Knowledge from this project will facilitate and inform our decisions about individual patients undergoing pharmacological treatment.

DETAILED DESCRIPTION:
Acetylcholinesterase inhibitors (AChE-I) comprise the major class of drugs used to treat Alzheimer's disease (AD). Despite widespread use, there is controversy about the usefulness of these medications. Concerns have been modest response rates of treated versus placebo groups, relatively small effect sizes with respect to efficacy, drug costs, and clinical relevance of the effects. One problem is that measures of efficacy used may not be sufficiently sensitive to detect a true drug effect. Another problem is that changes noted after 4-6 months of therapy confound the drug effect and the natural progression of the disease. Lastly, patient heterogeneity may contribute to the wide range of degree of response, further decreasing overall effect sizes. The investigators address three important issues to improve the clinical usefulness of cholinergic therapy. First, outcome measures are needed that are sensitive to the effects of cholinergic treatment. Second, outcome measures should be sensitive to the drug effect early in the course of treatment before a measurable decline of the disease progression occurs. Third, improved treatment would be attained if specific patient characteristics or performance measures were identified, which contributed to, or even predicted who will likely benefit. The premise of the current proposal is that measures of higher-order attention - currently omitted from standard assessments of treatment outcome - can provide insight into early efficacy of cholinergic treatment. The investigators are conducting a preliminary study that supports our hypotheses by testing the value of such attentional measures. The rationale for using attentional measures is as follows: (1) Attentional deficits are recognized as a critical cognitive change in the earliest phases of AD; (2) Attentional function, particularly tasks that tax available attentional capacity, is mediated by the cholinergic system; and (3) Acetylcholine is depleted in AD. However, the link between attention and cholinergic depletion in AD has not been fully explored, particularly with regard to response to cholinergic treatment. Surprisingly, attentional measures have not been included in the evaluation of AChE-I in the treatment of AD. The investigators propose that attentional performance could serve as a highly sensitive outcome measure and a marker of response.

Study aims and hypotheses

1. To determine that higher-order attentional measures are sensitive to the effect of cholinergic change early in the course of treatment. The investigators predict that performance on attentional tasks will improve in AChE-I treated patients compared to placebo controls after 7±1 weeks of treatment.

2. 2a. To examine the effect of cholinergic treatment on attentional measures as compared with global measures or measures of other cognitive domains. The investigators predict that the performance on tasks of attention is more sensitive than traditional global measures of performance.

2b. To examine whether cholinergic treatment changes the relationships among measures of attention and measures of other cognitive function. The prediction is that that the relationships among attention and cognitive domain measures will change with treatment.

3. To determine whether performance at 7±1 weeks can predict response at 6 months 3a. Patient response to AChE-I may be influenced by demographic variables, or influence performance in one or more cognitive domains. The aim is to determine which cognitive domain or demographic characteristic best predicts treatment response at six months. It is hypothesized that attention and memory (both mediated by cholinergic mechanisms) will best predict treatment response seen at six months.

3b. To determine whether an attentional change seen in patients early in the treatment course predicts drug response. It is hypothesized that change in attention measured between baseline and 7±1 weeks will predict overall improvement in those patients who show positive treatment response at six months.

Knowledge gained from this project will facilitate and inform our decisions about individual patients undergoing pharmacological treatment. The application of these goals can apply to current AChE-I treatment as well as other treatments, such as those now involving combined cholinergic and glutaminergic agents.

BACKGROUND AND SIGNIFICANCE Attention and Alzheimer's disease (AD): The vulnerability of higher-order attention tasks in AD occurs in tasks such as selective attention, and covert orienting. Attentional deficits are documented in patients with prodromal AD who later develop the disease, suggesting potential sensitivity of attention to disease onset. Mechanisms of attention are mediated via anterior executive control (required in conjunctive search and inhibitory control) and via posterior disengagement. The deficits in AD may be explained by regional frontal or posterior dysfunction, or by a disconnection between the frontal and posterior attentional networks that disrupt the feedback system. Acetylcholine and attention: A primary modulator of attention is acetylcholine (ACh). Decreased ACh impairs attentional function in animals and humans including vigilance in rat, covert orienting in primate and AD, and complex attention in human airplane pilots. ACh functions in a dose related manner, with increased task load of higher background noise correlating with increased ACh release. Cholinergic antagonists (e.g., scopolamine) slow reaction time (RT) and increase omission errors on visual search, and increase omission and commission errors on signal detection. Higher scopolamine doses slow RT in covert orienting in primates involving inferior parietal regions.

AD, attention and cholinesterase inhibitors: The relationship between attention and acetylcholine has not been well demonstrated in the assessment of AChE-I. Efficacy studies of donepezil, galantamine or rivastigmine show modest effect sizes ranging from 1.8-4.1 points on the 70 point Alzheimer Disease Assessment Scale - Cognitive section (ADAS-Cog) scale. These small effect sizes may partially be a function of using this outcome measure, which obscures the sensitivity to attention and memory with a global score. Targeted cognitive domains may be better response indicators. In a post-mortem analysis of AD patients, regions of low cholinergic activity correlated to memory and attention.

Moreover, after 12 weeks of galantamine treatment, AD patients who reached therapeutic dose showed faster RT, better choice reaction time and in memory, recognition of faces. Also, on functional imaging, early response to AChE-I appears to affect regions that mediate directed attention.

In summary, if attentional function is intrinsically linked to the level of cholinergic activity, it should used be an outcome measure of AChE-I treatment in AD to improve treatment sensitivity.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of Alzheimer's Disease
* Mini Mental State Examination score >15 / 30
* Can swallow pills

Exclusion Criteria:

* No other dementia due to Parkinson's disease, Lewy Body dementia, Normal Pressure Hydrocephalus, Fronto-temporal dementia, or prominent cerebral vascular accident
* No prior or concurrent use of cholinesterase inhibitors
* No prior or concurrent use of memantine hydrochloride
* No other concurrent anticholinergic treatments

Ages: 50 Years to 95 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2005-12-01 (Actual); Primary Completion 2009-07-31 (Actual); Study Completion 2021-01-13 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nancy Foldi, PhD, Principal Investigator — NYU Winthrop Hospital
Locations (1):
- Winthrop-University Hospital, Mineola, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Vila-Castelar C, Ly JJ, Kaplan L, Van Dyk K, Berger JT, Macina LO, Stewart JL, Foldi NS. Attention Measures of Accuracy, Variability, and Fatigue Detect Early Response to Donepezil in Alzheimer's Disease: A Randomized, Double-blind, Placebo-Controlled Pilot Trial. Arch Clin Neuropsychol. 2019 May 1;34(3):277-289. doi: 10.1093/arclin/acy032. PMID 29635383

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Of 25 individuals enrolled, 2 participants allocated to the placebo group discontinued: one complained of side-effects (n = 1); one moved from NY area (n = 1). Total N= 23.
Groups:
- Placebo: Participants in the placebo group first received oral administration of a placebo pill for approximately 6 weeks. After that initial interval, the study was unblinded and participants in the placebo group then received 5mg of donepezil hydrochloride treatment for 6 months.
  The Placebo group was evaluated at baseline, after 6 weeks of placebo, after 6 weeks of donepezil hydrochloride drug treatment, and 6 months of donepezil hydrochloride treatment.
  Donepezil Hydrochloride: 5mg of Donepezil Hydrochloride by mouth
  Placebo: prepared placebo looking exactly the same as drug. Participants took placebo by mouth for approximately 6 weeks, and after unblinding, they took donepezil hydrochloride for 6 months.
Period: Overall Study
Arm/Group | Drug | Placebo
Started | 12 | 11
Completed | 12 | 11
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Drug | Placebo | Total
Number analyzed (Participants) | 12 | 11 | 23
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 12 | 11 | 23
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 8 | 7 | 15
  Male | 4 | 4 | 8
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 12 | 11 | 23
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 23
Mini Mental State Examination (MMSE) [Mean (Standard Deviation); unit: units on a scale] — Mini Mental Status Examination (MMSE). Points generated range from 0 - 30, with higher score indicating better performance. There are no subscale scores. Scores of 25-30 can be considered within norm, and <25 indicate cognitive impairment. Reference: Folstein, M. F., Folstein, S. E., & McHugh, P. R. (1975). Mini-Mental State: A practical method for grading the cognitive state of patients for the clinician. Journal of Psychiatric Research, 12, 189-198. doi:0022-3956(75)90026-6 [pii]
  units on a scale | 24.3 (3.5) | 25.4 (1.7) | 24.9 (2.6)
Dementia Rating Scale (DRS) [Mean (Standard Deviation); unit: units on a scale] — Standard measure used in Geriatric Clinical settings. Points generated testing domains of Attention and Initiation&Perseveration; Construction; Conceptuatlization; and Memory. Total possible points = 144; Below 130 indication of presence of dementia Mattis, S. (1988). Dementia Rating Scale: Professional Manual. Odessa, FL: Psychological Assessment Resources, Inc.
  0-144 score; higher is better
  units on a scale | 119.7 (10.4) | 127.1 (7.2) | 123.4 (8.8)
Clinical Dementia Rating Scale (CDRS) [Mean (Standard Deviation); unit: units on a scale] — This standard measure is widely used in dementia research. Sum of Box scores are used to rank degree of perceived functional and memory and functional impairment ranging from 0 - 6: 0 is considered within norm; 0.5 mild impairment; any score equal to or greater than 1.0 and up to 6.0 indicates increasing impairment.
  This is a global measure, assessed by judgment of the examiner and discussion with caregiver; it does not specify distinct cognitive domains. Morris, J. C. (1993). The clinical dementia rating scale (CDR): Current version and scoring rules. Neurology, 43(11), 2412-2414.
  units on a scale | 1 (.4) | 3 (.4) | 1.9 (.41)
Geriatric Depression Scale (GDS) [Mean (Standard Deviation); unit: units on a scale] — This measure assesses degree of Depressive symptomatology, developed and normed for the geriatric population. Range of possible scores from 0 - 30 points with cutoff points as follows: normal-0-9; mild depression; 10-19; severe depression -20-30. [reference: Yesavage, J., Brink TL, Rose T, et al. Development and validation of a geriatric depression screening scale: a preliminary report. Journal of Psychiatric Research, 1983;17 (1):37-49.]
  units on a scale | 6.7 (6.2) | 6.5 (4.5) | 6.6 (5.4)
Neuropsychiatric Inventory (NPI) [Mean (Standard Deviation); unit: units on a scale] — Neuropsychiatric Inventory; Cummings et al, Neurology 1994; 44:2308-2314), a validated informant-based interview that assesses neuropsychiatric symptoms over the previous month on frequency and severity of behaviors. range of point scores = 0 - 144 points, where lower score is better
  units on a scale | 16.7 (12.3) | 15.4 (15.8) | 16.1 (14.1)
ADAS- Cog [Mean (Standard Deviation); unit: units on a scale] — This Alzheimer's Disease Assessment Scale-Cognitive Subscale (ADAS-Cog) remains primary metric for drug efficacy. The possible score range from 0 to 70 summing the number of errors made all tasks: higher scores indicate worse performance.
  Rosen, W. G., Mohs, R. C., & Davis, K. L. (1984). A new rating scale for Alzheimer's disease. American Journal of Psychiatry, 141, 1356-1364.
  units on a scale | 17.3 (6.6) | 13.1 (3.8) | 15.2 (5.2)
HVLT Learning [Mean (Standard Deviation); unit: units on a scale] — A list of 12 nouns with four words drawn from each of three semantic categories is read to participant .Scores are derived for Total Recall after learning trials, Delayed Recall, and % Retention and a Recognition Discrimination based on yes/no questions from a list of 24 words (12 original words, 6 distractors from the same semantic categories 6 unrelated distractors. Discrimination index' (cut-off score 19) can be obtained. Scoring : 0-36 total words recalled, higher score is better.
  units on a scale | 11 (2.6) | 11.4 (3.8) | 11.2 (3.2)
HVLT delay Recall [Mean (Standard Deviation); unit: units on a scale] — see description of Hopkins Verbal Learning Test at Learning. For this delayed recall score, rang of abilities is 0(low)-12 (high) words recalled; scores range from 0-12, higher score is better.
  units on a scale | 1.2 (1) | 1.1 (1.4) | 1.1 (1.2)
HVLT Recognition [Mean (Standard Deviation); unit: units on a scale] — see description of Hopkins Verbal Learning Test at Learning. Scores range from 0-12 indicating the number of words recognized after a delay, higher score is better.
  units on a scale | 5.3 (3.6) | 6.7 (2.7) | 6.0 (3.15)
Letter Fluency [Mean (Standard Deviation); unit: units on a scale] — Ability to generate words starting with a letter (e.g., F, A or S). One minute for each letter. Total score is number of correct words for each letter with no points for repetitions, non-words, proper nouns or names. Score is the maximum items generated; ranging from 0 (low) - indefinite, higher score is better.
  units on a scale | 9.0 (5.0) | 9.4 (4.3) | 9.2 (4.6)
Category Fluency [Mean (Standard Deviation); unit: units on a scale] — Ability to generate words from three different categories (e.g., fruits, vegetables and animals within a minute for each category. Total score is number of correct words for each category with no points for repetitions or non-words. score range 0 to unlimited, where 0 = low score, higher score is better.
  units on a scale | 7.4 (2.7) | 7.9 (2.7) | 7.5 (2.7)
Visual Form Discrimination [Mean (Standard Deviation); unit: units on a scale] — Visual Form Discrimination, Arthur L. Benton, PhD. Visual non-verbal tests designed as a convenient procedure to assess the capacity for complex visual form discrimination. Maximum score = 32. range 0-32; 32 max accuracy score, higher score is better.
  units on a scale | 26.7 (3.9) | 27.9 (2.5) | 27.3 (3.2)
Digit Span Forward (max) [Mean (Standard Deviation); unit: units on a scale] — Participants are asked to repeat series of numbers in same order as given by the examiner. Scoring is based on the quantity of numbers recited. Maximum numbers reached is the participant's best forward digit score. Scores range from 0-9, higher score is better.
  units on a scale | 5.9 (0.9) | 6.0 (0.8) | 5.9 (0.8)
Digit Span Backward (max) [Mean (Standard Deviation); unit: units on a scale] — Participants are asked to repeat series of numbers in the reverse order as given by the examiner. Maximum numbers reached is the participant's best backward digit score of quantity of numbers recited. Scores range from 0-8, higher score is better.
  units on a scale | 3.6 (0.8) | 6.0 (0.8) | 4.8 (0.8)
DKEFS Trail Making Test-4 [Mean (Standard Deviation); unit: units on a scale] — "The D-KEFS Trail Subtest 4: Number-Letter Switching Scaled Score was used to assess executive functioning. Scaled scores range from 1-19. Higher scores represent less impairment (below 8 = low; 8-12 = average; > 12 = above average)".
  units on a scale | 12.2 (11.7) | 6.7 (6.2) | 9.5 (8.9)
DKEFS Trail Making Test-5 [Mean (Standard Deviation); unit: units on a scale] — Delis-Kaplan Executive Functions Test (D-KEFs) Trails - condition 5 was used to measure speed. Scaled scores range from 0-20 with higher scores seconds representing better performance.
  units on a scale | 62.7 (36.5) | 54.3 (16.6) | 58.5 (26.6)

OUTCOME MEASURES:

1. Primary Outcome: Change in Foreperiod Effect Task - Processing Speed
Description: Computerized attention task measures response time to detect a target presented at varied interstimulus intervals (350ms and 500ms). Participants respond to centrally presented asterisk on computer screen. Time elapsed from prior stimulus (= interstimulus interval) indicates when prior stimulus was presented. xx
Time Frame: Baseline to 6 weeks
Measure: Median (Standard Deviation); unit: response time in msec
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 11
response time in msec
  350 | 42 (176.3) | 13 (9)
  500 | 33 (176.7) | 13 (9)

2. Primary Outcome: Change in Covert Orienting Task
Description: Computerized attention task measuring response time to detect a target after a spatial orienting cues of either valid (cue on same side in space as target) or Invalid Cue (cue on opposite side of space as target). Longer response time (msec) indicates worse performance.
Time Frame: Baseline to 6 weeks
Measure: Median (Inter-Quartile Range); unit: milliseconds
Groups:
- Drug: treatment group
- Placebo: placebo group
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 11 | 12
milliseconds | 496.5 [414.6 to 578.4] | 452.5 [401.7 to 503.3]

3. Primary Outcome: Change in Attentional Blink Task Baseline to 6 Weeks - Stimulus Onset Asynchrony (SOA) 266ms
Description: Computerized attention task measures the accuracy of reporting stimuli presented at time intervals, varying load. Faster reaction time and accuracy represents better performance.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Groups:
- Drug Treatment: All Participants received Donepezil Hydrochloride daily for 6 weeks.
  Donepezil Hydrochloride: 5mg of Donepezil Hydrochloride by mouth
Arm/Group | Drug Treatment
Number analyzed (Participants) | 23
milliseconds | -.06 (.32)

4. Primary Outcome: Change in Attentional Blink Task Baseline to 6 Weeks - SOA 399ms
Description: Computerized attention task measures the accuracy of reporting stimuli presented within 399 ms interval. Higher accuracy represents better performance.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: milliseconds
Arm/Group | Drug Treatment
Number analyzed (Participants) | 23
milliseconds | -.022 (.33)

5. Primary Outcome: Change of ADAS-COG From Baseline to 6 Months
Description: Change of Alzheimer's Disease Assessment Scale - Cognitive subscale (ADAS-Cog); primary outcome measure of drug efficacy. Minimum value = 0, maximum value = 70. Higher scores represent worse cognitive functioning.
Time Frame: Baseline to 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Drug Treatment: All Participants received Donepezil Hydrochloride daily for 6 months.
  Donepezil Hydrochloride: 5mg of Donepezil Hydrochloride by mouth
Arm/Group | Drug Treatment
Number analyzed (Participants) | 23
units on a scale | -.29 (4.70)

6. Primary Outcome: Foreperiod Effect Task at 6 Weeks - Fatigue (Blocks 1 & 2)
Description: Computerized attention task measures reaction time (RT) to detect a target presented at varied interstimulus interval comparing Block 1 (presented at beginning of session) and Block 2 (presented at end of session)
Time Frame: 6 weeks
Measure: Median (Standard Deviation); unit: msec
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 11
msec
  Block 1 | 400 (87.4) | 331 (200.7)
  Block 2 | 395 (85.3) | 385 (254.2)

7. Primary Outcome: Change in Foreperiod Effect Task - Variability (350ms & 500ms)
Description: Computerized attention task measures the variability (SD) in response time to detect a target presented at varied interstimulus intervals (350ms and 500ms)
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: msec
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 10
msec
  350ms | -26.7 (42.97) | -4.5 (34.44)
  500ms | 28.46 (110.63) | 8.37 (39.73)

8. Primary Outcome: Covert Orienting at 6 Weeks - Fatigue Across Blocks
Description: Computerized attention task measures response time to detect a target across blocks of stimuli. Data shown for performance at Block1 and Block5
Time Frame: 6 weeks
Measure: Median (Standard Deviation); unit: msec
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 11
msec
  Block 1 | 415 (145.1) | 402 (95.1)
  Block 5 | 451 (134.2) | 487 (144.3)

9. Primary Outcome: Neuropsychiatric Inventory Score
Description: Neuropsychiatric Inventory (NPI) is a scale that measures neuropsychiatric symptoms. We reported a score that captures the frequency of each symptom multiplied by the severity rating score. Scores range from 0 - 144; Higher scores represent worse outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug Treatment
Number analyzed (Participants) | 23
score on a scale | 14.09 (14.26)

10. Secondary Outcome: Change in Dementia Rating Scale
Description: Dementia Rating Scale (DRS) change score (performance at 6 weeks minus performance at baseline). This is a global measure of cognitive function. Scores range from 0 - 144; higher scores represent better cognitive functioning.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 11
units on a scale | 1.67 (6.91) | -.54 (6.27)

11. Secondary Outcome: Mini Mental Status Examination
Description: Mini Mental Status Examination (MMSE) is a commonly used cognitive screener. Scores range from 0-30; higher scores mean better cognitive functioning.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 10
units on a scale | -.17 (2.44) | -1.09 (2.02)

12. Secondary Outcome: Alzheimer's Disease Assessment Scale - Cognitive (ADAS-Cog)
Description: as for outcome 5
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 10
score on a scale | -1.90 (4.92) | .99 (2.25)

13. Secondary Outcome: Change in Digit Span Forward
Description: This measure represents the change in the variable longest Digit Span Forward (LDSF) from baseline to 6 weeks. Score represents the maximum length of number repeated in the forward condition. Score ranges from 0 to 9. Higher scores represent better outcome.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 10
units on a scale | -0.6 (1) | -0.4 (0.75)

14. Secondary Outcome: Change in Hopkins Verbal Learning Test- Revised - Recall
Description: Hopkins Verbal Learning Test- Revised (HVLT-R) (Brandt, 1991) is a list-learning task. Recall variable is computed by adding the number of words repeated in each of the three learning trials. Raw scores of each measure were used in the analyses. Total Recall ranges from 0-30. Higher scores represent better outcome.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 10
score on a scale | .17 (1.8) | .40 (4.79)

15. Secondary Outcome: Change in Language Function Assessed With the Letter Fluency Test
Description: Letter fluency (FAS) (Benton, 1967) was selected to assess speed of verbal generativity. Participants are required to generate words that start with a particular letter (excluding n; three trials (words starting with 'F', 'A', 'S' each for 1 minute minutes) are administered. Higher performance is better with range from 0 to unlimited.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Drug: Participants in the Drug group received oral 5mg of Donepezil Hydrochloride daily for 6 months. The Drug group was assessed at baseline, after approximately 6 weeks. The baseline to 6 weeks phase was part of the double-blind, placebo controlled portion of the trial.
  Donepezil Hydrochloride: 5mg of Donepezil Hydrochloride by mouth
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 9
score on a scale | .003 (1.51) | .17 (2.52)

16. Secondary Outcome: Change on Trail Making Test - Condition
Description: The Delis-Kaplan Executive Function (D-KEFS Trail) Subtest 4: Number-Letter Switching Scaled Score was used to assess executive functioning. Scaled scores range from 1-19. Higher scores represent less impairment (below 8 = low; 8-12 = average; > 12 = above average). Scores represent seconds to complete the task. Faster performance is better.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 10
units on a scale | -1.67 (39.45) | -2.3 (41.46)

17. Secondary Outcome: Change in Visual Form Discrimination
Description: Measure of visuospatial function requiring matching designs from the Benton Visual Form Discrimination test. Total scores is calculated by adding the number of items correct. Total score ranges from 0-32, higher score is better.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 11
score on a scale | .92 (3.09) | .33 (3.94)

18. Secondary Outcome: Change in Category Fluency Test
Description: Measure of language / semantic function. This task requires participants to generate words belonging to specific categories within 1 minute. There are three trials. Total scores is computed by obtaining the mean number of words generated across the three trials (fruits/vegetables/animals). Higher score represents better outcome.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 10
score on a scale | .17 (5.56) | -2.8 (4.02)

19. Primary Outcome: Instrumental Activities of Daily Living
Description: Scale of instrumental activities of daily living (IADLs), adapted from Lawton Brody scale. Caregiver rates 8 functional items from 0-2 severity. Total score is the sum of ratings for each item. Total score ranges from 0 (minimum) to 16 (maximum) with higher scores representing worse functional outcomes.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug Treatment
Number analyzed (Participants) | 23
units on a scale | 6.54 (4.23)

20. Secondary Outcome: Change in Digit Span Backwards
Description: This measure represents the change in the variable longest Digit Span Backwards (LDSB) from baseline to 6 weeks. Score represents the maximum length of number repeated in the backward condition. Score ranges from 0 to 8. Higher scores represent better outcome.
Time Frame: Baseline to 6 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Drug | Placebo
Number analyzed (Participants) | 12 | 10
units on a scale | 0.5 (0.8) | 0.1 (0.75)

ADVERSE EVENTS:
Time Frame: 6 Months
Arm/Group | Drug | Placebo
All-Cause Mortality (participants affected / at risk) | 0/12 | 0/11
Serious Adverse Events (participants affected / at risk) | 0/12 | 0/11
Other Adverse Events (participants affected / at risk) | 0/12 | 0/11

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2006-09-07): https://cdn.clinicaltrials.gov/large-docs/76/NCT03073876/Prot_SAP_000.pdf